CLINICAL TRIAL: NCT07091604
Title: Objective Skin Pigmentation Assessment in Healthy Volunteers and in Patients With Skin Disease: An Observational Study Using Non-invasive Skin Imaging
Brief Title: An Observational Study to Assess Objective Skin Pigmentation Variation.
Acronym: SKIN-IMAGING
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, dmwbalak, Principal Investigator, Leiden University Medical Center
Other Study IDs: NL-009794
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Skin Diseases; Healthy Skin
Keywords: Skin pigmentation; Melanin index; Colorimetry; Multispectral imaging; Line-Field Confocal Optical Coherence Tomography; Skin parameters; Skin colour; Skin color; Etnicity; TEWL; Erythema index; Non-invasieve measurement; Skin Disease; Skin of Colour; Laser speckle contrast imaging
MeSH Terms: conditions — Skin Diseases; Pigmentation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy volunteers with diverse skin tones
- Patients: Any patient with a skin condition under treatment by a dermatologist with active lesions.

SUMMARY:
Accurate assessment of skin pigmentation is essential in dermatology for properly diagnosing and managing a wide range of skin conditions. Traditionally, skin colour has been evaluated through visual inspection or by using classifications like the Fitzpatrick skin type. However, these methods can be subjective, culturally biased, and often are centered around lighter skin tones, which may lead to misdiagnosis or inappropriate treatment for individuals with darker skin.

With advances in technology, non-invasive imaging tools such as colorimetry and multispectral imaging now offer more precise and objective ways to measure skin pigmentation. These methods can help provide consistent and unbiased information about skin tone, benefiting both clinical care and research. Despite these technological advances, there is currently no agreed-upon standard for how to measure skin pigmentation objectively in everyday clinical practice or research settings.

This study aims to explore better, more accurate ways to measure skin pigmentation using modern, non-invasive imaging technologies. Traditional methods for assessing skin colour, like visual inspection or classifying by ethnicity, are often unreliable and biased. In this study, researchers will use tools such as colorimetry and multispectral imaging to measure skin pigmentation more objectively.

The study includes two groups of participants: healthy adults and adults with skin conditions. Researchers will measure a value called the melanin index, which reflects the amount of pigment in the skin, and compare it across different areas of the body and among people with different skin tones and conditions.

The goal is to understand how skin pigmentation varies and to see if these new technologies can help doctors more accurately diagnose and manage skin diseases for people of all skin types.

ELIGIBILITY:
Inclusion Criteria:-

* Age ≥ 18 years
* Ability to understand oral and written Dutch or English

Exclusion Criteria:

For study cohort #1 (Healthy volunteers):

* Extensive tattoos covering >50% of the total body area
* Recent extensive sun exposure (e.g. sun tanning booth or stay in a tropical country) in the last 3 weeks
* Use of self-tanner products in the last 3 weeks

For study cohort #2 (Patients):

* Extensive tattoos covering >50% of the total body area
* Extensive skin lesions covering >50% of the total body area
* Recent extensive sun exposure (e.g. sun tanning booth or stay in a tropical country) in the last 3 weeks
* Use of self-tanner products in the last 3 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For study cohort #1 (healthy volunteers): adult subjects will be recruited at multiple locations to ensure a diverse study population reflecting the full spectrum of skin colour types. Firstly, volunteers will be recruited using flyers at the campus of Leiden University. Along with that, partners of patients visiting the outpatient dermatology clinic of the LUMC. Lastly, subjects will be asked to partake in the study at public spaces (e.g. museums, festivals) that have given consent for this. Thus, subjects will be recruited in person by researchers at the aforementioned sites, through physical advertisements and digital advertisements.
  For study cohort #2 (patients with any skin disease): adult subjects with be recruited at the outpatient dermatology clinic of the LUMC and the affiliated hospitals of the CONNECTED (Clinical Network for Trials in Dermatology) in the Randstad region (e.g., The Hague, Zoetermeer, and Amsterdam).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-07-22 (Estimated); Primary Completion 2027-01-22 (Estimated); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
Melanin index | At baseline study visit (single time point)
  Melanin index as measured by skin colorimetry and multispectral imaging.

SECONDARY OUTCOMES:
Fitzpatrick skin type | At baseline study visit (single time point)
  Self-questionnaire and assessed by dermatologist
Age | At baseline study visit (single time point)
Ethnicity | At baseline study visit (single time point)
  Self-reported
Line-Field Confocal Optical Coherence Tomography (LC-OCT) | At baseline study visit (single time point)
  LC-OCT is a non-invasive optical imaging technique based on a combination of the optical principles of optical coherence tomography and reflectance confocal microscopy with line-field illumination, which can generate cell-resolved images of the skin, in vivo, in vertical section, horizontal section and in three dimensions.
3D Multispectral imaging | At baseline study visit (single time point)
  The redness, melanin and superficial morphology of (non-)lesional skin sites and healthy skin will be determined using a 3D multispectral imaging system.
Colorimetry | At baseline study visit (single time point)
  The melanin, redness and surface characteristics of (non-)lesional and healthy skin will be assessed using a colorimetry device that quantitatively measures skin color parameters, including melanin, based on reflected light.
Skin barrier function by Skin Barrier Pro | At baseline study visit (single time point)
  The barrier status by trans epidermal water loss of (non-)lesional skin and healthy skin will be determined using Skin Barrier Pro
VISIA | At baseline study visit (single time point)
  VISIA is a non-invasive imaging system designed for in vivo analysis of facial skin, utilizing multi-spectral imaging and digital analysis to assess various skin features, including pigmentation, porphyrins, texture, and wrinkles. The system captures standardized, high-resolution images under different lighting conditions (including cross-polarized and UV light), allowing for both surface and subsurface visualization of the skin. It provides quantitative and comparative assessments of skin health and damage, supporting both clinical evaluation and cosmetic or dermatological research.
Patient and Observer Scar Assessment Scale | At baseline study visit (single time point)
  POSAS is a validated scar assessment tool that combines both patient-reported outcomes and clinical evaluation to provide a comprehensive assessment of scar quality. It consists of two complementary parts: the Observer Scale, completed by a clinician, which evaluates vascularity, pigmentation, thickness, relief, pliability, and surface area; and the Patient Scale, completed by the individual, which captures subjective symptoms such as pain, itching, and overall opinion of the scar. POSAS enables standardized, semi-quantitative scoring of scars, facilitating both clinical monitoring and research on scar treatment outcomes.
Laser speckle contrast imaging | At baseline study visit (single time point)
  Laser speckle contrast imaging (LSCI) is a non-invasive optical imaging technique used to assess microvascular blood flow in vivo by analyzing the speckle pattern produced when coherent laser light is scattered by moving red blood cells. The resulting speckle contrast is inversely related to the velocity of blood flow, enabling real-time, high-resolution visualization of perfusion over large skin areas without the need for contrast agents. LSCI is particularly suited for dynamic monitoring of vascular responses in dermatology, wound healing, and inflammatory skin conditions.
Scarletred® Vision | At baseline study visit (single time point)
  Scarletred® Vision is a digital, non-invasive skin imaging and analysis platform that enables objective and standardized quantification of skin conditions over time using smartphone-based photography combined with a calibrated color patch and proprietary software. The system captures high-resolution images under controlled lighting conditions and applies automated analysis algorithms to quantify parameters such as erythema, pigmentation, and lesion area. By providing reproducible, color-calibrated data, Scarletred® Vision supports longitudinal skin monitoring in clinical trials and dermatological research, including evaluation of treatment effects in inflammatory and pigmentary disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided